CLINICAL TRIAL: NCT06613035
Title: Twice-per-week Selinexor, 2 Days Melphalan Plus BU2FLU3 Compared with BU3FLU5 for Elder High-risk Acute Myeloid Leukemia Undergoing Allogenic Hematopoietic Cell Transplantation: a Multi-center Randomized Phase 3 Trial
Brief Title: Twice-per-weekSelinexor, 2 Days Melphalan
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024062
Record Dates: First submitted 2024-09-22; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Acute Myeloid Leukemia
Keywords: allogeneic hematopoietic stem cell transplantation
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — selinexor; Melphalan; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SMBF group will receive the following Sel2Mel2BU2FLU3 conditioning regimen (Experimental): * Selinexor: 60 mg/day from days -9 to -5.
  * Melphalan: 60 mg/m² on days -8 and -7.
  * Intravenous Busulfan (Bu): 3.2 mg/kg on days -6 and -5.
  * Fludarabine (Flu): 30 mg/m² on days -4, -3, and -2.
  Interventions: Drug: Selinexor; Drug: Melphalan; Drug: Intravenous Busulfan; Drug: Fludarabine
- Patients in the BF group will receive the BU3FLU5 conditioning regimen (Experimental): * Intravenous Busulfan (Bu): 3.2 mg/kg on days -9, -8, and -7.
  * Fludarabine (Flu): 30 mg/m² on days -6, -5, -4, -3, and -2.
  Interventions: Drug: Intravenous Busulfan; Drug: Fludarabine

INTERVENTIONS:
Drug: Selinexor — Selinexor: 60 mg/day from days -9 to -5.
  Arms: SMBF group will receive the following Sel2Mel2BU2FLU3 conditioning regimen
Drug: Melphalan — Selinexor: 60 mg/day from days -9 to -5.
  Arms: SMBF group will receive the following Sel2Mel2BU2FLU3 conditioning regimen
Drug: Intravenous Busulfan — 3.2 mg/kg on days
Drug: Fludarabine — 30 mg/m² on days

SUMMARY:
Twice-per-week Selinexor, 2 days Melphalan plus BU2FLU3 compared with BU3FLU5 for elder high-risk acute myeloid leukemia undergoing allogenic hematopoietic cell transplantation: a multi-center randomized phase 3 trial

DETAILED DESCRIPTION:
Twice-per-week Selinexor, 2 days Melphalan plus BU2FLU3 compared with BU3FLU5 for elder high-risk acute myeloid leukemia undergoing allogenic hematopoietic cell transplantation: a multi-center randomized phase 3 trial Primary Objective The primary objective of this study is to compared 1-year RFS between Sel2Mel2BU2FLU3 and BU3FLU5 groups for elder AML in CRc undergoing allo-HCT.

Secondary Objective The secondary objective of this study is to compare leukemia relapse, engraftment, GVHD, OS, TRM, AEs and RRT between Sel2Mel2BU2FLU3 and BU3FLU5 groups

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with high-risk acute myeloid leukemia (excluding acute promyelocytic leukemia).

  2. Recipients of allogeneic hematopoietic stem cell transplantation (including HLA-matched or mismatched allogeneic transplantation as well as unrelated donor transplantation).

  3. Age ≥ 55 years. 4. Disease status prior to allogeneic transplantation must be complete remission (CRc), confirmed by bone marrow analysis within three days prior to randomization.

  5. Karnofsky Performance Score (KPS) of at least 60. 6. Informed consent must be signed prior to the commencement of the study procedures. If the patient's signature would be detrimental to their treatment due to their medical condition, the informed consent may be signed by a legal guardian or an immediate family member of the patient.

Note: *High-risk AML: ① Patients classified as high-risk according to the ELN 2022 grading criteria. ② AML patients with persistent MRD positivity prior to transplantation. ③ Patients with refractory or relapsed AML.

Exclusion Criteria:

* 1. Previous history of hematopoietic stem cell transplantation. 2. Active cardiac disease, defined as one or more of the following:

  1. History of uncontrolled or symptomatic angina.
  2. Myocardial infarction within the last 6 months prior to study enrollment.
  3. History of arrhythmias requiring medication or with clinically significant symptoms.
  4. Uncontrolled or symptomatic congestive heart failure (NYHA class > 2).
  5. Ejection fraction below the lower limit of the normal range. 3. Respiratory failure (PaO2 ≤ 60 mmHg). 4. Liver dysfunction (total bilirubin ≥ 3 mg/dL, transaminases > twice the upper limit of normal).

  5. Renal dysfunction (creatinine clearance rate < 30 mL/min). 6. Presence of psychiatric disorders or other conditions that prevent cooperation with the study treatment and monitoring requirements.

  7. ECOG performance status of ≥ 4. 8. Uncontrolled or active infection. 9. Any condition that impairs the ability to provide informed consent. 10. Any conditions deemed unsuitable for enrollment by the investigator prior to randomization.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
1-year RFS | 1-year
  The primary objective of this study is to compared 1-year RFS between Sel2Mel2BU2FLU3 and BU3FLU5 groups for elder AML in CRc undergoing allo-HCT.

SECONDARY OUTCOMES:
1-year OS | 1-year
  1-year OS
1-year GVHD | 1-year
  1-year GVHD

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Hebei Medical University Second Hospital, Shijiazhuang, Hebeisheng
  - Zhengzhou University First Affiliated Hospital, Zhengzhou, Henan
  - The 960th Hospital of the Joint Service Support Force of the Chinese People's Liberation Army, Jinan, Shandong
  - People's Liberation Army The General Hospital of Western Theater Command, Chengdu, Sichuan